CLINICAL TRIAL: NCT04590378
Title: Evaluation of the Patients With COVID-19 in Terms of Pulmonary Embolism
Brief Title: Pulmonary Embolism and COVID-19
Acronym: COVID-19-PE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Other Study IDs: UU-PE001
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Covid-19; Pulmonary Embolism
MeSH Terms: conditions — COVID-19; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 Patients with Pulmonary embolism: Clinically demonstared cases infected with COVID-19 who developed pulmonary embolism.
  Interventions: Other: intensive care unit admission ratio
- Covid-19 Patients without Pulmonary embolism: Clinically demonstared cases infected with COVID-19 who did not develop pulmonary embolism.
  Interventions: Other: intensive care unit admission ratio

INTERVENTIONS:
Other: intensive care unit admission ratio — intensive care unit admission ratio

SUMMARY:
The charts of patients who developed pulmonary embolism in the course of COVID-19 will be evaluated, retrospectively. Clinical features and laboratory data will be analyzed.

DETAILED DESCRIPTION:
Patients with COVID-19 infection will be evaluated retrospectively. Demographic data, clinical and laboratory findings will be recorded. Findings of patients with pulmonary embolism and withour pulmonary embolism will be compared.

ELIGIBILITY:
Inclusion Criteria:

- All patients with positive RT-PCR for COVID-19

Exclusion Criteria:

- All patients with negative RT-PCR for COVID-19

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All COVID-19 patients with positive RT-PCR tests will be analyzed retrospectively. Patients with and without pulmonary embolism will be compared in terms of age, gender, side disease, hospitalization in intensive care, mortality rates etc.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary embolism | 1 year
  development of pulmonary embolism

SECONDARY OUTCOMES:
Intensive care unit | 1 year
  need for admission to intensive care unit
mortality | 1 year
  mortality rate due to pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Cevdet Duran, M.D., Principal Investigator — Uşak University Medical School
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No